CLINICAL TRIAL: NCT05689567
Title: Effect of Peripheral Focus-out Glasses on Emmetropization in Chinese Children Aged 6-8 Years: 2 Years Randomized Clinical Trial.
Brief Title: Focus-out Glasses on Emmetropization in Chinese Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DEFOG
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Emmetropization; Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEFOG group (Experimental): Subjescts will wear DEFOG glasses(peripheral focus-out glasses).
  Interventions: Device: DEFOG glasses(peripheral focus-out glasses)
- Control group (No Intervention): Subjects in the control group will just be observed.

INTERVENTIONS:
Device: DEFOG glasses(peripheral focus-out glasses) — Subjects in the intervention group will wear peripheral focus-out glasses ≧8 hours a day and ≧5 days a week.
  Arms: DEFOG group

SUMMARY:
The purpose of this study is to characterize the effects of peripheral focous-out glasses on emmetropization in non-myopic Chinese Children Aged 6-8 Years.This is a prospective, parallel-controlled randomized trial.

DETAILED DESCRIPTION:
Myopia is one of the most common eye diseases that cause visual impairment and blindness, and the high rate of myopia in young people is a major public health issue. Based on the clinical studies of optical defocusing to regulate eye growth and refractive changes through visual signal feedback, we hypothesize that early wearing of peripheral defocus glasses in children can slow down the process of emmetropization and even prevent the onset of myopia by producing more myopic defocusing. The aim of this study is to investigate whether wearing peripheral defocus glasses can effectively delay emmetropization in non-myopic children aged 6-8 years , and to further explore its effect on preventing the onset of myopia.

The study adopts a 2-year，single-centre, randomized, parallel-controlled trial with a non-blinded design. Subjects who pass the screening period will have their baseline data collected and will be assigned to the experimental or control groups according to the randomization principle. The experimental group will be fitted with Direct Emmetropia with Focus-out Glasses (hereafter referred to as DEFOG) to guide the emmetropization process. The control group will be given no treatment and will be a blank control. Baseline data including visual acuity, cycloplegic objective refraction, axis length, accommodation amplitude, strabismus examination, pupil size, choroidal thickness and peripheral retinal refraction will be measured when enrolled in the group and follow-up data will be measured at month 6, 12, 18 and 24. The primary interest of this study will be studied by comparing the difference in cycloplegic objective refraction changes between month 24 and baseline in the two groups of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥6 and ≤8 years at enrollment.
2. At least one parent' s Spherical equivalent refraction≤-3.00D.
3. Spherical equivalent refractions (SERs) under cycloplegia: +0.50 to +1.50 diopters (D)
4. Astigmatism ≤1.00 D .
5. Anisometropia ≤1.00 D.
6. Best Corrected Visual Acuity (BCVA) : 1.0 or better
7. Provision of consent written by subject's legal guardian
8. Willing and able to participate in all required activities of the study

Exclusion Criteria:

1. Any of the following abnormalities on the ocular surface, such as trachoma, pemphigoid, chemical injury, heat burn, radiation injury, etc.
2. Eyelid abnormalities (e.g. entropion, ectropion, tumor, edema, blepharospasm, incomplete eyelid closure, severe trichiasis, severe ptosis) ,which affect eyelid function in either eye
3. Eye diseases such as strabismus, amblyopia, anisometropia, fundus diseases, and accommodation abnormality，etc.
4. Prior treatment of myopia control in either eye, including but not limited to drugs, orthokeratology, low-level red-light therapy, etc.
5. Noncompliance with measurement at enrollment.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Changes of Cycloplegic Objective Refraction(spherical equivalent refraction, SER)(D) | From baseline till the 24th month
  Changes of cycloplegic objective refraction(i.e reflected by SER) from baseline till the 24th month (only the right-eye data included). Objective refraction data will be examined by AUTO REF/KERATOMETER. Ciliary muscle paralysis will be performed by using 1% cyclopentanone eye drops, 2 doses in each eye, 2 doses 5 minutes apart. The optometry will be performed after 20 minutes of complete ciliary muscle paralysis (disappearance of pupil response to light or pupil diameter at least greater than 6 mm). SER is calculated by adding the sum of the sphere power with half of the cylinder power. Baseline data will be measured at the time of enrollment. Follow-up data will be measured on the 24th month from baseline. The 24th month data will be subtracted from the baseline data to obtain changes.

SECONDARY OUTCOMES:
Changes of Cycloplegic Objective Refraction(SER) (D) | The 6th month, the 12th month and the 18th month from baseline
  Changes of cycloplegic objective refraction (i.e reflected by SER) different follow-up time and the baseline time (only the right-eye data included). Objective refraction data will be examined by AUTO REF/KERATOMETER.
Cycloplegic Objective Refraction(SER)(D) | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Cycloplegic objective refraction (i.e reflected by SER) any follow-up time (only the right-eye data included). Objective refraction data will be examined by AUTO REF/KERATOMETER.
Myopia | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Cycloplegic SER≦-0.50D at any follow-up time. Objective refraction data will be examined by AUTO REF/KERATOMETER.
Changes of Axial Length(AL)(mm) | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Changes of Axial Length (AL) between different follow-up time and the baseline time (only the right-eye data included).AL will be examined by IOL Master.
Axial Length (AL) (mm) | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Axial Length (AL) at any follow-up time (only the right-eye data included).AL will be examined by IOL Master.
Amplitude of Accommodation (AMP)（D） | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Amplitude of Accommodation (AMP) at any follow-up time (only the right-eye data included). AMP will be examined by lens test.
Visual Acuity | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  The Logarithmic Visual Acuity at any follow-up time (only the right-eye data included).
Strabismus Examination（△） | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Strabismus examination at any follow-up time by SYNOPTOPHORE.
Changes of Choroidal Thickness (ChT) （um） | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Changes of Choroidal Thickness (ChT)between different follow-up time and the baseline time (only the right-eye data included). ChT will be examined by OPTICALCOHERENCETOMOGRAPHY.
Pupil size（mm） | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Pupil size at any follow-up time (only the right-eye data included).
Peripheral Retinal Refraction(D) | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Peripheral Retinal Refraction at any follow-up time (only the right-eye data included). Peripheral Retinal Refraction will be examined by AUTO FUNDUS CAMERA.
The percentage of participants with fast myopic shift | From baseline till the 24th month
  The percentage of participants with fast myopic shift over 2 years(only the right-eye data included). The fast myopic shift is defined as cycloplegic objective refraction (i.e reflected by SER) myopic shift of at least 1.00 D. Objective refraction data will be examined by AUTO REF/KERATOMETER.
Corneal curvature(D) or radius of curvature(mm) | The 6th month, the 12th month, the 18th month and the 24th month from baseline
  Corneal curvature or radius of curvature(only the right-eye included). They can be interconverted. Data will be examined by AUTO REF/KERATOMETER.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen L, He W, Yang W, Yan W, Yang C. Effect of wearing peripheral focus-out glasses on emmetropization in Chinese children aged 6-8 years: study protocol for a 2-year randomized controlled intervention trial. Trials. 2023 Nov 22;24(1):746. doi: 10.1186/s13063-023-07799-8. PMID 37993963